CLINICAL TRIAL: NCT03727399
Title: Identification of Allergen-reactive Antibodies in the Blood of Pollen Allergic Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Mabylon AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-01110
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pollen Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood withdrawal — Blood withdrawal

SUMMARY:
The project examines the hypothesis that monoclonal allergen-neutralizing antibodies can be recombinantly produced from B lymphocytes isolated from pollen allergic patients. Patient samples suitable for antibody cloning are selected based on seroprofiling for the respective allergens. The study aims at isolating lymphocytes from patients with potential allergen-neutralizing IgG in serum and to clone antibodies from antibody gene sequences obtained from B cells of those patients.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic rhinitis, conjunctivitis or asthma due to sensitization to grass- or birch Allergens
* Male or female patients older than 18 years
* Written informed consent for providing blood and also to allow experimental manipulation

Exclusion Criteria:

* Age < 18 years
* Any corticosteroids within the last three days
* Oral corticosteroid therapy within the last ten days
* Parenteral depot corticosteroids within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The project population will include adult (> 18 years) patients with a history of grass and birch pollen allergy verified by positive skin prick test and allergen-specific IgE in blood. The study population may also include patients with ongoing or completed AIT.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Antibody profiling | October 2018 - September 2021
  Analysis and IgG profiling of specific antibodies binding major grass- and tree-pollen allergens in allergic patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Immunologie Zentrum Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No